CLINICAL TRIAL: NCT05755633
Title: Role of Day +60 WT1 Assessment on Bone Marrow in Predicting Relapse and Mortality After Allogeneic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, CHIUSOLO PATRIZIA, PROFESSOR, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4065
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Assessment of the WT1 Expression Level on Bone Marrow Samples Collected at Day +60 After Allogeneic Stem

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The rationale of this study is to determine if an association exists between WT1 expression and relapse occurrence in patients with acute myeloid leukemia submitted to allogeneic stem cell transplantation. In particular, we want to studied WT1 expression level on bone marrow samples of day +60 in terms of predicting power on relapse incidence so as to determine a cut-off value for identify high risk patients.

DETAILED DESCRIPTION:
This is a retrospective study which will be held on 50 patients with acute myeloid leukemia allografted in the transplant Units of Policlinico Agostino Gemelli in Rome, between June 2018 and July 2020, for whom WT1 level was assessed on bone marrow at day 60 after transplant. The minimum follow up for surviving patients will be 60 days. Patients will be classified according to European Leukemia Net criteria. For each patient a total of 24 ml of bone marrow was collected at day +60 post transplant, whereas the same quantity of bone marrow was collected from healthy donor during bone marrow harvest procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years Diagnosis of acute myeloid leukemia Patients received allogeneic stem cell transplantation Signed informed consent to storage and use biological samples for research scope Signed informed consent to privacy

Exclusion Criteria:

* Patients who had received a previous stem cell transplant Hematological disease other than acute myeloid leukemia Patient not studied for WT1 level at day +60 after transplant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective study which will be held on 50 patients with acute myeloid leukemia allografted in the transplant Units of Policlinico Agostino Gemelli in Rome, between June 2018 and July 2020, for whom WT1 level was assessed on bone marrow at day 60 after transplant.
  The minimum follow up for surviving patients will be 60 days. Patients will be classified according to European Leukemia Net criteria
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
we want to studied WT1 expression level on bone marrow samples of day +60 in terms of predicting power on relapse incidence so as to determine a cut-off value for identify high risk patients | day 60 after transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Servizio E Dh Di Ematologia, Roma, Italy

IPD SHARING:
Plan to Share IPD: No